CLINICAL TRIAL: NCT02070926
Title: Coronary CT Angiography Evaluation for Clinical Outcomes in Asymptomatic Patients With Type 2 Diabetes Mellitus
Brief Title: The CRONOS-ADM Registry
Status: Completed | Type: Observational
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Kiyuk Chang, Associate professor, Seoul St. Mary's Hospital
Other Study IDs: ADM CCTA
Record Dates: First submitted 2014-02-23; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Asymptomatic Patients With Type 2 Diabetes Mellitus; Atherosclerosis; Coronary Artery Disease; Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years

GROUPS / COHORTS (2):
- Perform coronary CT angiography
- Do not perform coronary CT angiography

SUMMARY:
The CRONOS-ADM (Coronary CT angiography evaluation for clinical outcomes in asymptomatic patients with type 2 diabetes mellitus) registry is a large, prospective observational registry of demographic, clinical and laboratory data with long-term clinical outcome of asymptomatic diabetic patients without history of CAD or angina or angina-equivalent symptoms at two affiliated hospitals of The Catholic University of Korea.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Asymptomatic type 2 diabetes mellitus
3. Prospective data collection for CAD risk factors

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consist of patients with asymptomatic type 2 diabetes mellitus at two centers of catholic university of Korea
Sampling Method: Probability Sample
Dates: Start 2006-01; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Time to major adverse events | up to median 3 years follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee EY, Yang HK, Lee J, Kang B, Yang Y, Lee SH, Ko SH, Ahn YB, Cha BY, Yoon KH, Cho JH. Triglyceride glucose index, a marker of insulin resistance, is associated with coronary artery stenosis in asymptomatic subjects with type 2 diabetes. Lipids Health Dis. 2016 Sep 15;15(1):155. doi: 10.1186/s12944-016-0324-2. PMID 27633375